CLINICAL TRIAL: NCT00660153
Title: A Phase 1b, Open-Label, Dose-Escalation Study of Tivozanib (AV-951) Plus FOLFOX6 in Subjects With Advanced Colorectal Cancer and Other Gastrointestinal Cancers
Brief Title: Study of Tivozanib (AV-951) Plus FOLFOX6 in Subjects With Advanced Colorectal Cancer and Other Gastrointestinal Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-951-103
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Colorectal Cancer; Gastrointestinal Cancer
Keywords: Advanced Colorectal Cancer and Other Gastrointestinal Cancers; tivozanib; AV-951
MeSH Terms: conditions — Colorectal Neoplasms; Gastrointestinal Neoplasms | interventions — tivozanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm; multiple cohort (Experimental): Single arm; multiple cohort
  Interventions: Drug: Tivozanib (AV-951) plus FOLFOX6

INTERVENTIONS:
Drug: Tivozanib (AV-951) plus FOLFOX6 — Investigational product, dosage and mode of administration (1 cycle = 4 weeks of treatment):
  Tivozanib (AV-951): 0.5 mg, 1.0 mg, and 1.5 mg oral once daily On Day -5 (± 2 days) subjects will receive a single dose of tivozanib (AV-951) for pharmacokinetic sampling. Beginning on Day 1 of Cycle 1, subjects will receive tivozanib (AV-951) once daily for 3 weeks followed by 1 week off. Tivozanib (AV-951) dosing repeats every cycle in the absence of disease progression or unacceptable toxicity. On days when both tivozanib (AV-951) and the FOLFOX6 chemotherapy regimen are co-administered, tivozanib (AV-951) will be administered immediately prior to the start of the FOLFOX6 chemotherapy regimen.
  Subjects will receive FOLFOX6 chemotherapy every 2 weeks starting on Day 1 of Cycle 1. Subjects will receive 2 treatments of FOLFOX6 in each treatment cycle, starting on Day 1 and Day 15.

SUMMARY:
The FOLFOX6 regimen is a standard chemotherapy regimen for the treatment of patients with colorectal cancer and other gastrointestinal cancers. Tivozanib (AV-951) is a targeted anti-angiogenesis agent that has demonstrated acceptable tolerability in a phase I clinical trial. This study is designed to test the hypothesis that tivozanib (AV-951) can be combined with standard FOLFOX6 chemotherapy for the treatment of patients with colorectal and other gastrointestinal cancers. The purpose of this study is to determine the maximum dose of tivozanib (AV-951) that can be safely combined with FOLFOX6 chemotherapy, and to evaluate the safety profile, tolerability, and pharmacokinetics of this combination.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, study design that will examine safety, tolerability, and maximum tolerated dose of tivozanib (AV-951) and FOLFOX6 in advanced colorectal cancer and other gastrointestinal cancers. In the study, only the doses of tivozanib (AV-951) will be escalated from 0.5 mg/day to 1.5 mg/day. All subjects will receive standard doses of FOLFOX6 chemotherapy every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18-year-old males or females
2. Histologically or cytologically confirmed metastatic colorectal cancer or other gastrointestinal malignancy for which FOLFOX6 chemotherapy is a standard treatment. Other gastrointestinal cancers include, but are not limited to, esophageal, gastric, and small intestine, appendiceal, and pancreatico-biliary cancers.
3. Documented progressive disease
4. Measurable or evaluable disease by RECIST. (Note: Subjects enrolled in the MTD Expansion Cohort are required to have measurable disease, according to RECIST.)
5. No more than 2 prior chemotherapy regimens for metastatic disease (This does not include prior adjuvant chemotherapy with fluorouracil and/or oxaliplatin.)
6. At least 3 weeks since prior treatment with:

   * Chemotherapy (at least 6 weeks for nitrosoureas, mitomycin C, and liposomal doxorubicin)
   * Agents targeting the VEGF pathway (eg, bevacizumab, sunitinib, sorafenib, etc.)
   * Other signal transduction inhibitors and monoclonal antibodies
   * Immunotherapy or biological response modifiers
   * Systemic hormonal anti-cancer therapy, with the exception of LHRH agonists for prostate cancer
   * Any experimental therapy
7. Resolution of toxicities associated with prior chemotherapy to ≤ Grade 1 (except for Grade 2 alopecia)
8. ECOG performance status ≤ 2 (see Appendix A) and life expectancy ≥ 3 months
9. No childbearing potential or use of effective contraception by all fertile male and female subjects during the study and for 30 days after the last dose of study drug. All subjects must agree to use a highly effective method of contraception (including their partner). Effective birth control includes (a) IUD plus one barrier method; or (b) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
10. Dated and signed informed consent

Exclusion Criteria:

1. Primary CNS malignancies or clinically active CNS metastases
2. Hematologic malignancies (includes leukemia in any form, lymphoma, and multiple myeloma)
3. Any of the following hematologic abnormalities:

   * Hemoglobin < 9.0 g/dL
   * ANC < 1500 per mm3
   * Platelet count < 100,000 per mm3
4. Any of the following serum chemistry abnormalities:

   * Total bilirubin > 1.5 × ULN
   * AST or ALT > 2.5 × ULN (or > 5 x ULN for subjects with liver metastasis)
   * GGT > 2.5 x ULN (or > 5 x ULN for subjects with liver metastasis)
   * Alkaline Phosphatase > 2.5 x ULN (or > 5 x ULN for subjects with liver or bone metastasis)
   * Serum albumin < 3.0 g/dL
   * Creatinine > 1.5 × ULN (or calculated CLCR <50 mL/min/1.73 m2)
   * Proteinuria > 2.5 g/24 hours or 3+ with urine dipstick
   * Any other ≥ Grade 3 laboratory abnormality at baseline (other than those listed above)
5. Significant cardiovascular disease, including:

   * Active clinically symptomatic left ventricular failure
   * Active HTN (diastolic blood pressure > 100 mmHg). Subjects with a history of hypertension must have been on stable doses of anti-hypertensive drugs for ≥ 4 weeks prior to start of Cycle 1
   * Uncontrolled hypertension: Blood pressure >140/90 mmHg on more than 2 antihypertensive medications
   * Myocardial infarction within 3 months prior to start of Cycle 1
6. Serious/active infection, or infection requiring parenteral antibiotics
7. Inadequate recovery from any prior surgical procedure or major surgical procedure within 6 weeks prior to the start of Cycle 1
8. Unhealed wounds, ulcers, or bone fractures
9. Ongoing hemoptysis or history of clinically significant bleeding
10. Cerebrovascular accident within 12 months prior to the start of Cycle 1, or peripheral vascular disease with claudication on walking less than 1 block
11. Deep venous thrombosis or pulmonary embolus within 12 months prior to the start of Cycle 1 and/or ongoing need for full-dose oral or parenteral anticoagulation
12. History of ≥ Grade 3 hypersensitivity reaction with prior exposure to oxaliplatin
13. Subjects with a "currently active" second malignancy other than non-melanoma skin cancers or localized prostate cancer (with stable PSA for at least 3 months prior to the start of Cycle 1). Subjects are not considered to have a "currently active" malignancy if they have completed anti-cancer therapy and are considered by their physician to be a < 30% risk of relapse.
14. Life-threatening illness or organ system dysfunction compromising safety evaluation
15. Uncontrolled psychiatric disorder or altered mental status precluding informed consent or necessary testing
16. Inability to comply with protocol requirements
17. Pregnant or lactating women
18. Known concomitant genetic or acquired immune suppression disease, such as HIV
19. Consumption of herbal preparations/supplements (except for a daily multivitamin/mineral supplement not containing herbal components) within 2 weeks prior to the start of Cycle 1
20. Prior radiotherapy:

    * Local radiation therapy (involving ≤ 25% of bone marrow) within 2 weeks prior to the start of Cycle 1
    * Craniospinal radiotherapy within 3 months prior to the start of Cycle 1
    * Radiotherapy to: whole abdomen or pelvis, whole lungs, > 25% of bone marrow, or total body irradiation within 6 months prior to the start of Cycle 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability, and maximum tolerated dose of tivozanib (AV-951) in combination with FOLFOX6 chemotherapy. | • Minimum of 4 weeks for assessment of tolerability, minimum of 8 weeks (2 consecutive dosing cycles) for assessment of anti-tumor activity. Extended therapy may continue for up to 1 year from the subject's start of Cycle 1.

SECONDARY OUTCOMES:
To characterize the pharmacokinetic profile of tivozanib (AV-951) and FOLFOX6 chemotherapy when administered together, and to assess the antineoplastic activity of the combination of tivozanib (AV-951) and FOLFOX6 chemotherapy. | • Minimum of 4 weeks for assessment of tolerability, minimum of 8 weeks (2 consecutive dosing cycles) for assessment of anti-tumor activity. Extended therapy may continue for up to 1 year from the subject's start of Cycle 1.

CONTACTS AND LOCATIONS:
Overall Officials: Ferry Eskens, MD, PhD, Principal Investigator — Erasmus Medical Center; Department of Medical Oncology; E.G.E de Vries, Prof, MD, Principal Investigator — University Medical Center Groningen; Jaroslow Jac, MD, Study Director — AVEO Pharmaceuticals, Inc.
Locations (2):
- Netherlands (2):
  - University Medical Center Groningen; Internal Medicine, Department of Medical Oncology, Groningen
  - Erasmus Medical Center; Department of Medical Oncology, Rotterdam

REFERENCES:
- [Derived] Oldenhuis CN, Loos WJ, Esteves B, van Doorn L, Cotreau MM, Strahs AL, den Hollander MW, Gietema JA, de Vries EG, Eskens FA. A phase Ib study of the VEGF receptor tyrosine kinase inhibitor tivozanib and modified FOLFOX-6 in patients with advanced gastrointestinal malignancies. Clin Colorectal Cancer. 2015 Mar;14(1):18-24.e1. doi: 10.1016/j.clcc.2014.12.001. Epub 2014 Dec 16. PMID 25591799